CLINICAL TRIAL: NCT02855619
Title: Comparison of the Incidence of 3 Inspiratory Muscle Training Programs on Inspiratory Strength, on Difficult to Wean Patients in Intensive Care Unit: a Multi-centre Randomised Trial.
Brief Title: Comparison of the Impact of Three Programs of Inspiratory Muscles.
Acronym: PREDRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2015/25
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: inspiratory muscles training programs; Ventilator-induced diaphragmatic dysfunction; Weaning; Intensive care unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Martin (Active Comparator): A threshold-based IMT is performed like used by Martin in a randomized trial in 2011, in a view of inspiratory strength increase.
  Interventions: Procedure: Martin
- Cader (Active Comparator): A threshold-based IMT is performed like used by Cader in a randomized trial in 2012, in a view of inspiratory endurance increase.
  Interventions: Procedure: Cader
- EDRIC (Experimental): A new threshold-based IMT is performed, in a view of both inspiratory strength and endurance increase.
  Interventions: Procedure: EDRIC

INTERVENTIONS:
Procedure: Martin — The physiotherapist perform the IMT using the threshold IMT inspiratory muscle trainer, connected to the intubation tube. He manage the resistance to the higher resistance tolerated by the patient in a set of 6 breaths. Participant repeats 4 sets of 6-10 breaths with 2 minutes of resting with mechanical ventilation between each set.
  This treatment is made twice a day, 7days per week from inclusion to extubation exept if Glasgow score is under 8, hyperthermia more than 39°c, haemodynamic's instability, or hypoxemia( PaO2/FiO2<150).
  Arms: Martin
Procedure: Cader — The physiotherapist perform the IMT using the threshold IMT inspiratory muscle trainer, connected to the intubation tube. He manage the resistance to 30% of the Maximal Inspiratory Pressure initially recorded the day of the inclusion. Participant breaths against this resistance during 5 minutes. The resistance is daily increased of 10 % to the higher tolerated.
  This treatment is made twice a day, 7days per week from inclusion to extubation exept if Glasgow score is under 8, hyperthermia more than 39°c, haemodynamic's instability, or hypoxemia( PaO2/FiO2<150).
  Arms: Cader
Procedure: EDRIC — The physiotherapist perform the IMT using the threshold IMT inspiratory muscle trainer, connected to the intubation tube. He manage the resistance at 30% of the Maximal Inspiratory Pressure of the day for the first set of 20 breaths with a resistance 's increasment of 10% at each set. Participant repeats 4 sets of 20 breaths with 2 minutes of resting with mechanical ventilation between each set.
  This treatment is made twice a day, 7days per week from inclusion to extubation exept if Glasgow score is under 8, hyperthermia more than 39°c, haemodynamic's instability, or hypoxemia( PaO2/FiO2<150).
  Arms: EDRIC

SUMMARY:
Ventilator-induced diaphragmatic dysfunction appears to contribute to slow weaning from mechanical ventilation. Several trials of inspiratory muscle training to facilitate weaning in intensive care have been performed, with inconsistent results, utilizing different methods of IMT in different populations.

In this study, the investigators want to compare the incidence of 3 inspiratory muscle training programs on inspiratory strength, on difficult to wean patients in intensive care unit.

This is a multi-center randomized trial not blinded with 3 parallels groups:

* Martin's group: a threshold-based IMT is performed like used by Martin in a randomized trial in 2011, in a view of inspiratory strength increase.
* Cader's group: a threshold-based IMT is performed like used by Cader in a randomized trial in 2010 , in a view of inspiratory endurance increase.
* EDRIC's group: a new treshold-based IMT is performed, in a view of both inspiratory strength and endurance increase.

The investigators think that a new threshold-based IMT performed in a view of both inspiratory strength and endurance increase, is more effective and well tolerated than the 2 others protocols.

DETAILED DESCRIPTION:
The main objective of this study is to determinate which IMT program is the most effective on the inspiratory muscle strength and endurance increase. The investigators will be able to study the impact on the weaning time of IMT performed with the best protocol.

The investigators are going to conduct a randomized trial with intention-to-treat analysis. Following 18h of invasive mechanical ventilation in a controlled mode, the failure of the first single breathe trial of 2 hours and the presence of sevrability criterias defined by the European consensus conference in 2007, 88 participants will be included. Participants will be randomizesd to receive one of the 3 protocols of IMT, 2 times per day, 7 days per week, from the inclusion to the extubation.

The ratio of randomization will be 1:1:2 for a better evaluation of EDRIC's group wich propose a new IMT protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient ventilated more than 18h in a controlled mode;
* First single breathe trial of 2 hours failure;
* Presence of sevrability criterias definied by the European consensus conference in 2007 an usually used:

  * diminution of the sedfative agents,
  * Patients with spontaneous beath in VAC mode or patient ventilated in a VSAI-PEP mode,
  * PaO2/FiO2 ≥150,
  * Absence d'inotropes ou de vasopresseurs à forte dose ou dose croissante (<1mg/h),
  * SaO2 > 90% with FiO2 ≤ 50%,
  * PEP ≤ 8cmH2O,
  * Corporal température between 36°C and 39°C,
  * Glasgow Score ≥ 8.

Exclusion Criteria:

* Age < 18 years ;
* medically unstable;
* Poor vital pronostic at very short term;
* Cardiac arrest with a poor neurological prognostic;
* Neuromuscular disease ;
* Pneumothorax non drained ;
* Tracheostomy ;
* Current pregnancy ;
* Patients with guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure score (inspiratory muscle strength index) performed by an external electronic device connected with a unidirectional valve. | Baseline and up to day 25

SECONDARY OUTCOMES:
Peak Pressure (inspiratory muscle endurance index) performed by an incremental threshold test. | Baseline and up to day 25
Duration of the weaning period | up to day 25
ICU lengh of stay | Day 30
Weaning success | up to day 27
Adverse events | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perez, Professor, Study Chair — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Réanimation Médicale, Bordeaux
  - Réanimation Médicale, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reginault T, Martinez Alejos R, Coueron R, Burle JF, Boyer A, Frison E, Vargas F. Impacts of three inspiratory muscle training programs on inspiratory muscles strength and endurance among intubated and mechanically ventilated patients with difficult weaning: a multicentre randomised controlled trial. J Intensive Care. 2024 Jul 25;12(1):28. doi: 10.1186/s40560-024-00741-3. PMID 39049092